CLINICAL TRIAL: NCT00122330
Title: Randomized, Double-Blind, and Placebo-Controlled Study Using Eculizumab in Transfusion Dependent PNH Patients
Brief Title: Study Using Eculizumab in Transfusion Dependent Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: TRIUMPH
Record Dates: First submitted 2005-07-18; First posted 2005-07-22 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Hemoglobinuria, Paroxysmal
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

INTERVENTIONS:
Drug: eculizumab

SUMMARY:
The primary objective is to evaluate the safety and efficacy of eculizumab in transfusion dependent patients with hemolytic PNH.

ELIGIBILITY:
Inclusion Criteria:

* Must have required at least 4 transfusions in the past 12 months
* PNH type III red blood cell (RBC) clone by flow cytometry of >10%
* Lactate dehydrogenase (LDH) level > 1.5 x upper limit of normal
* Platelet count > 100,000/mm3
* Patient taking erythropoietin must be on a stable dose for at least 26 weeks
* Patient taking immunosuppressants must be on a stable dose for at least 26 weeks
* Patient taking corticosteroids must be on a stable dose for at least 4 weeks
* Patient taking coumadin must be at a stable INR for at least 4 weeks
* Patient taking iron supplements or folic acid must be on a stable dose for 4 weeks
* Willing and able to give written informed consent
* Must avoid conception

Exclusion Criteria:

* Mean hemoglobin level prior to transfusion over the previous 12 months is >10.5 gm/dl
* Absolute neutrophil count <500/ul
* Active bacterial infection
* Hereditary complement deficiency
* Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedures within 30 days
* Pregnant, breast-feeding, or intending to conceive
* History of meningococcal disease
* History of bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2004-10; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (43):
- United States (16):
  - City of Hope National Medical Center, Div. of Hematology & Bone Marrow Transplant, Duarte, California
  - University of California at Los Angeles, Los Angeles, California
  - Scripps Cancer Center, San Diego, California
  - Stanford University Medical Center, Division of Hematology, Stanford, California
  - Hartford Hospital, Cancer Clinical Research Office, Hartford, Connecticut
  - Cleveland Clinic, Dept. of Clinical Research, Weston, Florida
  - Indiana University Cancer Pavilion, Div. of Hematology-Oncology, Hematological Malignancy Program/Immunology, Indianapolis, Indiana
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - National Heart, Blood, and Lung Institute, National Institutes of Health, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, Dept. of Internal Medicine/Division of Hematology, St Louis, Missouri
  - NYU Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Health System, Division of Cell Therapy, Heme Malignancies Program, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Presbyterian Medical Center, PENN Comprehensive Hemophilia & Thrombosis Program, Philadelphia, Pennsylvania
- Australia (4):
  - Princess Alexandra Hospital, Oncology Haematology Radiation Department, Woolloongabba, Queensland
  - Queen Elizabeth Hospital, Dept. of Haematology, Woodville South, South Australia
  - Royal Melbourne Hospital, Dept. of Clinical Haematology & Medical Oncology, Parkville, Victoria
  - The Royal Perth Hosptial, Department of Haematology/Level 2, Perth, Western Australia
- Ucl St. Luc, Hematology Department, Brussels, Belgium
- University of Alberta, Cross Cancer Institute, Edmonton, Alberta, Canada
- France (2):
  - Hospital De L'Hotel Dieu, Hematologie et Oncologie Medicale, Cedex, Paris
  - Hopital Saint-Louis, Centre G. Hayem-Secteur Bleu Porte 7, Laboratoire De Pathologie/Greffe de Moelle, Cedex, Paris
- Germany (5):
  - Universitatsklinikum Essen, Zentrum fur Innere Medizin, Essen
  - Universitatsklinik Greifswald, Innere Medizin C - Hamato-Onkologie, Greifswald
  - Medizinische Hochschule Hannover, Abt. Hamatologie/Onkologie, Zentrum fur Innere Medizin, Hanover
  - Saarland University Medical School, Internal Medicine 1, Homburg/Saar
  - Institut fur Klinische Transfusionmedizin und Immungenetik, Abtlg. Transfusionsmedizin des Universitatskinikums Ulm, Ulm
- St. James Hospital, Haematology Department, Dublin, Ireland
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Dipartimento di area critica medico-chirurgica, Florence
  - Ospedale San Martino, Dept. of Hematology, Genova
  - Ospedale Maggiore di Milano, Divisione di Ematologia, Milan
  - Universitar degli Studi di Napoli, Divisione di Ematologia, Azienda Universitar Policlinico, Napoli
  - Ospedale San Bortolo, Divisione di Ematologia, Vicenza
- UMC St. Radboud, Dept. of Hematology, Nijmegen, GA, Netherlands
- Sweden (2):
  - Lund University Hospital, Department of Internal Medicine, Section of Hematology, Lund
  - Umea University Hospital, Dept. of Internal Medicine 3, Section for Hematology, Umeå
- Universitatsklinik Basel, Division of Hematology, Basel, CH, Switzerland
- United Kingdom (4):
  - Royal Cornwall Hospital, Haematology Dept., Truro, Cornwall
  - Belfast City Hospital, Dept. of Haematology C Floor, Belfast
  - Leeds General Infirmary, D Floor Brotherton Wing, Leeds
  - St. George's Hospital, Department of Haematology, London

REFERENCES:
- [Result] Hillmen P, Young NS, Schubert J, Brodsky RA, Socie G, Muus P, Roth A, Szer J, Elebute MO, Nakamura R, Browne P, Risitano AM, Hill A, Schrezenmeier H, Fu CL, Maciejewski J, Rollins SA, Mojcik CF, Rother RP, Luzzatto L. The complement inhibitor eculizumab in paroxysmal nocturnal hemoglobinuria. N Engl J Med. 2006 Sep 21;355(12):1233-43. doi: 10.1056/NEJMoa061648. PMID 16990386
- [Derived] Hill A, Rother RP, Wang X, Morris SM Jr, Quinn-Senger K, Kelly R, Richards SJ, Bessler M, Bell L, Hillmen P, Gladwin MT. Effect of eculizumab on haemolysis-associated nitric oxide depletion, dyspnoea, and measures of pulmonary hypertension in patients with paroxysmal nocturnal haemoglobinuria. Br J Haematol. 2010 May;149(3):414-25. doi: 10.1111/j.1365-2141.2010.08096.x. Epub 2010 Mar 8. PMID 20230403